CLINICAL TRIAL: NCT00033267
Title: A Phase II Study of CCI-779 in Previously Treated Patients With Mantle Cell Non-Hodgkin's Lymphoma
Brief Title: CCI-779 in Treating Patients With Mantle Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01870; NCI-2012-01870 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCCTG-N0186; CDR0000069269; N0186 (Other: North Central Cancer Treatment Group); N0186 (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — temsirolimus; Sirolimus

ARMS (1):
- Treatment (Experimental): Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with stable disease receive a maximum of 6 courses. Patients with partial response receive a maximum of 12 courses. Patients with CR receive 2 additional courses beyond CR.
  Interventions: Drug: temsirolimus

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel

SUMMARY:
Phase II trial to study the effectiveness of CCI-779 in treating patients who have mantle cell non-Hodgkin's lymphoma. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the objective responses in patients with previously treated mantle cell non-Hodgkin's lymphoma treated with CCI-779.

II. Determine the toxic effects of this drug in these patients. III. Determine whether this drug inhibits cell proliferation pathways in these patients.

OUTLINE:

Patients receive CCI-779 IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with stable disease receive a maximum of 6 courses. Patients with partial response receive a maximum of 12 courses. Patients with complete response (CR) receive 2 additional courses beyond CR.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed mantle cell non-Hodgkin's lymphoma (MCL)
* Relapsed, refractory, or stable disease after prior chemotherapy, radiotherapy, or immunotherapy
* Unidimensionally measurable lymph node or lesion

  * At least 2.0 cm by CT scan or MRI OR at least 1.5 cm by physical exam
  * One of the following measurement parameters may be used:

    * Splenic enlargement may be used as a measurement parameter if spleen is palpable at least 3.0 cm across left costal margin
    * Malignant lymphocytosis may be used as a measurement parameter if absolute lymphocyte count is at least 5,000/mm^3
* No known CNS involvement (parenchymal mass or leptomeningeal involvement)
* Performance status - ECOG 0-2
* At least 3 months
* See Disease Characteristics
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 8 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Direct bilirubin ≤ 1.5 times ULN
* AST ≤ 3 times ULN (5 times ULN if liver metastases are present)
* Creatinine ≤ 2 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Cholesterol ≤ 350 mg/dL
* Triglycerides ≤ 400 mg/dL
* HIV negative
* No other active malignancy requiring treatment or that would preclude study participation
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* See Disease Characteristics
* Prior high-dose therapy with stem cell transplantation allowed
* At least 7 days since prior immunotherapy or other non-myelosuppressive biologic response modifiers
* See Disease Characteristics
* See Biologic therapy
* At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy for MCL
* Concurrent corticosteroids for adrenal insufficiency allowed
* See Disease Characteristics
* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy for MCL
* Any number of prior treatments allowed
* No other concurrent investigational or commercial agents for MCL
* No concurrent drugs that induce cytochrome p450 (e.g., carbamazepine, phenobarbital, phenytoin, ketoconazole, diltiazem, rifampin, terfenadine, cisapride, astemizole, or pimozide)
* No concurrent immunosuppressive therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-04; Primary Completion 2006-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve a confirmed CR or PR during the first 24 weeks of treatment defined by the International Workshop criteria | Up to 24 weeks
  The proportion will be evaluated separately for each dose group. The proportion of patients who achieve a confirmed CR or PR, or success, will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Time to progression | Time from registration to the time of progression, assessed up to 5 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Overall survival | Time from registration to death due to any cause, assessed up to 5 years
  The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Progression-free survival | Time from registration to progression or death due to any cause, assessed up to 5 years
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Duration of response | From the date of study registration until the date of progression in the subset of patients who respond, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ansell, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States